CLINICAL TRIAL: NCT04321681
Title: Diaphragm Ultrasound to Predict Posteroperative Residual Blockade
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jie YI, deputy director of surgery department, Peking Union Medical College Hospital
Other Study IDs: DiaphragmUltra
Record Dates: First submitted 2020-03-18; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Ultrasonography; Residual Curarization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study is a prospective observational research approved by the Ethics Committee of the Peking Union medical college Hospital. Patients scheduled for elective non-abdominal and non-thoracic surgery among age of 19-65 years and American Society of Anesthesiologists Physical Status Classification(ASA) I or II were inrolled. Diaphragm ultrasonogram was measured pre and post operation. Diaphragm excursion and diaphragm thickening fraction during quiet breathing as well as deep breathing were assessed. Neuromuscular monitor was performed during operation, after proper calibration.

ELIGIBILITY:
Enrollment criteria：

1. Patients who were scheduled for elective non-abdominal and non-thoracic surgery in Peking Union medical college hospital.
2. age of 19-65 years
3. American Society of Anesthesiologists Physical Status Classification(ASA) I or II.
4. Agree to informed consent

Exclusion criteria ： Patients with neuromuscular diseases, diaphragmatic palsy, thoracic malformation, hand disabilities, chronic obstructive pulmonary disease, severe liver or kidney diseases, electrolyte or acid-base disorders, morbid obesity (body mass index ≥30 kg/m2), pregnancy, allergy to drugs used in the study, use of medication interfering neuromuscular transmission within 72hours and patients with predicted difficulty in maintenance of airway were excluded from this study. Written informed consent will be obtained before preoperative evaluation by an anesthesiologist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective non-abdominal and non-thoracic surgery in Peking Union medical college hospital. All were among age of 19-65 years and American Society of Anesthesiologists Physical Status Classification(ASA) I or II.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
TOFr at extubation | within1 min before extubation
  Neuromuscular function was monitored thoughout operation based neuromuscular monitoring guideline by an independent investigator. TOF ratio before extubation was recorded. The scale of TOFr range from 0 to 1. TOFr<0.9 indicate existance of residual neuromuscular blockade.
Diaphragm ultrasound parameter | within 1 min after extubation
  Diaphragm excursion and thickening fraction was measured through ultrasonography within 2 min after extubation. Correlation between TOFr ratio and diaphragm parameters was explored.

SECONDARY OUTCOMES:
reintubation rate | within 24 hour
  If patients cannot breath by themselves after extubation, They need to be reintubated and mechanical ventilation need to be use to sustain their breathing.
Posteroperative pulmonary complication | 1 month
  incidence of airway obstruction, bronchospasm, pulmonary aspiration of gastric contents, apnea, unexpected ICU admissions, atelectasis and pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China